CLINICAL TRIAL: NCT02289209
Title: A Phase II Trial of Reirradiation Combined With Open Label Pembrolizumab in Patients With Locoregional Inoperable Recurrence or Second Primary Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Reirradiation With Pembrolizumab in Locoregional Inoperable Recurrence or Second Primary Squamous Cell CA of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dan Zandberg (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Dan Zandberg, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 18-009
Record Dates: First submitted 2014-10-17; First posted 2014-11-13 (Estimated); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Recurrent Head and Neck Cancer; Carcinoma, Squamous Cell of Head and Neck
Keywords: head and neck cancer; reirradiation; MK-3475; Anti-PD-1 monoclonal antibody; Squamous cell carcinoma; Keytruda; pembrolizumab
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — Re-Irradiation; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Reirradiation + MK-3475 (Experimental): Reirradiation 1.2 Gy BID for 5 days a week for 5 weeks with MK-3475 (Keytruda, pembrolizumab) 200mg intravenous every 3 weeks until 3 months post completion of reirradiation.
  Interventions: Radiation: Reirradiation; Drug: MK-3475

INTERVENTIONS:
Radiation: Reirradiation — Reirradiation 1.2 GY BID 5 days a week for 5 weeks.
Drug: MK-3475 — MK-3475 will be given at 200mg intravenous every 3 weeks starting day one of reirradiation and will be continued once every 3 weeks until 3 months post completion of reirradiation. Further continuation of MK-3475 will be determined by response evaluation at 3 months post completion of reirradiation
  Other Names: Keytruda, pembrolizumab

SUMMARY:
Eligible participants with locoregional inoperable recurrence or second primary squamous cell carcinoma of the head and neck will be treated with reirradiation combined with anti-PD-1 mAb MK-3475 (generic name: pembrolizumab, trade name Keytruda®).

DETAILED DESCRIPTION:
Each participant will undergo screening and then be treated with reirradiation with 1.2 Gy BID, 5 days a week (weeks 1-5). MK-3475 (generic name: pembrolizumab, trade name Keytruda®) will be given at 200mg intravenous every 3 weeks starting day one of reirradiation and will be continued in all participants until 3 months post completion of reirradiation, at which time a PET/CT will be done to evaluate response. Participants with progressive disease (PD) will be taken off MK-3475 and followed for survival. Participants that have a complete response (CR) will be followed clinically and radiographically, and if disease recurs may be eligible to be retreated with MK-3475 for up to one year. Participants with partial response (PR) or stable disease (SD) will continue treatment with MK-3475 for up to two years unless one of the following occurs:

* documented disease progression
* unacceptable adverse event(s)
* intercurrent illness that prevents further administration of treatment
* investigator decision to withdraw the subject
* withdrawal of consent
* pregnancy
* noncompliance
* administrative reasons (i.e. trial is closed prematurely).

Participants who have not progressed at completion of 24 months of therapy will be observed, but may be eligible for 1 year of retreatment with MK-3475 if they develop recurrence/progression and qualify for retreatment as detailed in the protocol,and if the trial is still ongoing.

ELIGIBILITY:
Patients with biopsy proven locoregional recurrence or second primary SCCHN which is unresectable or the patient is unwilling to undergo resection. Determination of unresectability will be based on multidisciplinary review of each case.

Inclusion Criteria:

1. Have received only prior radiation treatment course. Prior radiation course must have been with curative intent.
2. At least 6 months since completion of radiation
3. Based on prior radiation records, have had most of the tumor volume (>50%) previously radiated at doses > 45 Gy without exceeding spinal cord tolerance (combining previous and future radiation dose to spinal cord of < 50 Gy).
4. Be willing to undergo percutaneous endoscopic gastrostomy (PEG) placement, if necessary.
5. Have at least one measurable area of disease based on RECIST 1.1 within the previously radiated field.
6. Have provided adequate tissue for PD-L1 analysis either from an archival tissue sample or fresh biopsy done to confirm recurrence/second primary. Archival tissue sample can only be used if done within 3 months of enrollment on the clinical trial.
7. Performance status of 0 or 1 on the ECOG Performance Scale.
8. Life expectancy greater than 12 weeks
9. Adequate organ function as defined by the protocol

Exclusion Criteria:

1. Presence of distant metastatic disease.
2. Is currently participating in or has participated in a study of an investigational agent or used an investigational device within 4 weeks of the first dose of treatment.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has had a prior monoclonal antibody, chemotherapy, or targeted small molecule therapy within 4 weeks prior to study Day 1 or who has not recovered from adverse events due to agents administered more than 4 weeks earlier.
5. History of other malignancy within 5 years with the exception of prior Squamous cell carcinoma of the head and neck, adequately treated basal cell or squamous cell skin cancer, or carcinoma of the cervix.
6. Has an active autoimmune disease
7. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
8. Has an active infection requiring systemic therapy
9. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
10. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
11. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
12. Has received a live vaccine within 30 days prior to the first dose of trial treatment
13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Zandberg, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (4):
- United States (4):
  - Univeristy of Maryland - Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reirradiation + MK-3475
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Reirradiation + MK-3475
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.17 (8.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Number of months from the date of initiation of treatment to the date of progression of disease or death (whichever occurs first). Progressive disease, per RECIST 1.1, is defined as: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 36 months (after starting reirradiation and MK-3475)
Population: All treated patients who were radiologically evaluable and experienced disease progression.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Reirradiation + MK-3475
Number analyzed (Participants) | 48
months | 7.9 [4.3 to 10.2]

2. Secondary Outcome: Best Overall Response Rate (ORR)
Description: The percentage of the patients who have either Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm, or, Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. The patient's best overall response rate defined as the best response recorded from the start of the treatment until disease progression will be recorded, per RECIST 1.1.
Time Frame: Up to 36 months (after initiation of treatment with reirradiation and MK-3475)
Population: All treated patients who achieved radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Reirradiation + MK-3475
Number analyzed (Participants) | 23
percentage of patients | 56.1 [39.7 to 71.95]

3. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: The percentage of patients that have achieved a complete response, partial response, and stable disease as defined by RECIST 1.1. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm, Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters, or Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Up to 36 months (after initiation of treatment with reirradiation and MK-3475)
Population: All treated patients who achieved radiologic response or stable disease.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Reirradiation + MK-3475
Number analyzed (Participants) | 32
percentage of participants | 78.0 [62.4 to 89.4]

4. Secondary Outcome: Time to in Field Disease Progression
Description: Number of months from initiation of treatment to progression of disease within the radiation field.Progressive disease, per RECIST 1.1, is defined as: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 36 months (after initiation of treatment with reirradiation and MK-3475)
Population: Zero patients with results.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Reirradiation + MK-3475
Number analyzed (Participants) | 48
months | 13.1 [9.1 to NA] — Upper bound of 95% CI not reached due to low number of events.

5. Secondary Outcome: Overall Survival (OS)
Description: Number of months from first treatment until death. Patients who are alive will be censored at the last date of patient contact.
Time Frame: Up to 36 months (after initiation of treatment with reirradiation and MK-3475)
Population: All patients enrolled in the trial.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Reirradiation + MK-3475
Number analyzed (Participants) | 48
months | 13.1 [9.4 to 21.5]

6. Secondary Outcome: Quality of Life Using EORTC QLQ-C30 - Baseline
Description: Patient reported outcomes will be measured using EORTC QLQ-C30 questionnaires. This tool contains 30 items. It measures 5 functional dimensions (physical, role, cognitive, social, emotional), 6 single items (appetite loss, constipation, dyspnea, financial impact, sleep disturbance, diarrhea), 3 symptom items (fatigue, pain, nausea/vomiting) and a global health and quality of life scale. Scales range in score from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology or problems.
Time Frame: At Baseline
Population: Treated patients who completed Quality of Life evaluations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reirradiation + MK-3475
Number analyzed (Participants) | 48
score on a scale
  Global Health Status | 58.33 (24.06)
  Physical Functioning | 77.69 (24.55)
  Role Functioning | 66.33 (30.90)
  Emotional Functioning | 71.53 (26.06)
  Cognitive Functioning | 78.47 (25.02)
  Social Functioning | 66.67 (32.43)
  Fatigue | 36.34 (29.15)
  Nausea and Vomiting | 8.50 (16.36)
  Pain | 44.44 (32.86)
  Dyspnea | 13.61 (20.32)
  Insomnia | 34.69 (35.33)
  Appetite Loss | 23.61 (30.72)
  Constipation | 25.85 (32.82)
  Diarrhea | 10.20 (23.77)
  Financial concerns | 21.09 (30.95)

7. Secondary Outcome: Quality of Life Using EORTC QLQ-C30 - Cycle 3
Description: as for outcome 6
Time Frame: At Cycle 3 (Week 6)
Population: Treated patients who completed Quality of Life evaluations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reirradiation + MK-3475
Number analyzed (Participants) | 41
score on a scale
  Global Health Status | 59.96 (18.93)
  Physical Functioning | 78.37 (21.38)
  Role Functioning | 63.01 (32.81)
  Emotional Functioning | 81.25 (23.93)
  Cognitive Functioning | 76.83 (23.53)
  Social Functioning | 73.17 (29.32)
  Fatigue | 41.46 (28.33)
  Nausea and Vomiting | 10.57 (13.31)
  Pain | 41.67 (29.96)
  Dyspnea | 16.26 (22.51)
  Insomnia | 29.27 (30.91)
  Appetite Loss | 31.67 (32.86)
  Constipation | 19.51 (24.69)
  Diarrhea | 5.69 (14.72)
  Financial concerns | 15.45 (23.68)

8. Secondary Outcome: Quality of Life Using EORTC QLQ-C30 - Cycle 9
Description: as for outcome 6
Time Frame: At Cycle 9 (Week 26)
Population: Treated patients who completed Quality of Life evaluations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reirradiation + MK-3475
Number analyzed (Participants) | 25
score on a scale
  Global Health Status | 61.00 (24.26)
  Physical Functioning | 74.93 (30.57)
  Role Functioning | 64.00 (33.22)
  Emotional Functioning | 77.78 (24.16)
  Cognitive Functioning | 75.33 (33.03)
  Social Functioning | 71.33 (30.63)
  Fatigue | 40.00 (31.75)
  Nausea and Vomiting | 8.67 (21.58)
  Pain | 40.00 (37.27)
  Dyspnea | 9.33 (22.61)
  Insomnia | 29.33 (35.12)
  Appetite Loss | 19.44 (32.48)
  Constipation | 20.00 (30.43)
  Diarrhea | 4.00 (11.06)
  Financial concerns | 17.33 (30.61)

9. Secondary Outcome: Quality of Life Using EORTC QLQ-C30 - 12 Months
Description: as for outcome 6
Time Frame: At 12 months
Population: Treated patients who completed Quality of Life evaluations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reirradiation + MK-3475
Number analyzed (Participants) | 10
score on a scale
  Global Health Status | 72.50 (16.69)
  Physical Functioning | 84.67 (16.94)
  Role Functioning | 85.00 (16.57)
  Emotional Functioning | 85.00 (16.57)
  Cognitive Functioning | 91.67 (14.16)
  Social Functioning | 86.67 (23.31)
  Fatigue | 14.44 (17.41)
  Nausea and Vomiting | 0.00 (0.00)
  Pain | 26.67 (22.50)
  Dyspnea | 6.67 (21.08)
  Insomnia | 6.67 (21.08)
  Appetite Loss | 20.00 (23.31)
  Constipation | 3.33 (10.54)
  Diarrhea | 3.33 (10.54)
  Financial concerns | 16.67 (28.33)

10. Secondary Outcome: Quality of Life Using EORTC QLQ-C30 - 36 Months
Description: as for outcome 6
Time Frame: At 36 months
Population: Treated patients who completed Quality of Life evaluations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reirradiation + MK-3475
Number analyzed (Participants) | 3
score on a scale
  Global Health Status | 75.00 (22.05)
  Physical Functioning | 95.56 (3.85)
  Role Functioning | 88.89 (19.25)
  Emotional Functioning | 88.89 (12.73)
  Cognitive Functioning | 94.44 (9.62)
  Social Functioning | 66.67 (57.74)
  Fatigue | 11.11 (19.25)
  Nausea and Vomiting | 0.00 (0.00)
  Pain | 5.56 (9.62)
  Dyspnea | 0.00 (0.00)
  Insomnia | 11.11 (19.25)
  Appetite Loss | 11.11 (19.25)
  Constipation | 11.11 (19.25)
  Diarrhea | 0.00 (0.00)
  Financial concerns | 33.33 (57.74)

11. Secondary Outcome: Quality of Life Using EORTC QLQ-H&N 35 - Baseline
Description: Patient reported outcomes will be measured using the EORTC QLQ-H&N35, a 35-item questionnaire that assesses symptoms encountered specifically by patients with head and neck cancer. This measure generates 7 multiple-item scales (Pain, Swallowing, Senses, Speech, Social eating, Social contact, and Sexuality), in addition to 11 single items (eg, Opening mouth, Sticky saliva, Dry mouth, etc). Scales range in score from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology or problems.
Time Frame: At Baseline
Population: Treated patients who completed Quality of Life evaluations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reirradiation + MK-3475
Number analyzed (Participants) | 48
score on a scale
  Pain | 38.89 (33.21)
  Swallowing Problems | 40.08 (35.13)
  Sensory Problems | 32.58 (32.34)
  Speech Problems | 42.68 (31.69)
  Trouble with Social Eating | 39.07 (32.46)
  Trouble with Social Contact | 16.53 (20.07)
  Less Sexuality | 25.19 (37.54)
  Teeth Problems | 21.01 (36.08)
  Mouth Opening Problems | 48.61 (39.48)
  Dry Mouth | 46.53 (38.12)
  Sticky Saliva | 45.14 (42.66)
  Coughing | 35.46 (34.34)
  Feeling Ill | 27.08 (34.14)
  Painkiller Use | 74.47 (44.08)
  Nutritional Supplement Use | 62.50 (48.92)
  Feeding Tube Use | 37.50 (48.92)
  Weight Loss | 31.25 (46.84)
  Weight Gain | 20.83 (41.04)

12. Secondary Outcome: Quality of Life Using EORTC QLQ-H&N 35 - Cycle 3
Description: as for outcome 11
Time Frame: At Cycle 3 (Week 6)
Population: Treated patients who completed Quality of Life evaluations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reirradiation + MK-3475
Number analyzed (Participants) | 41
score on a scale
  Pain | 41.87 (32.09)
  Swallowing Problems | 45.83 (34.47)
  Sensory Problems | 43.24 (29.52)
  Speech Problems | 43.54 (27.89)
  Trouble with Social Eating | 47.97 (32.89)
  Trouble with Social Contact | 16.75 (23.79)
  Less Sexuality | 30.56 (39.14)
  Teeth Problems | 16.24 (29.49)
  Mouth Opening Problems | 54.47 (37.83)
  Dry Mouth | 51.22 (35.82)
  Sticky Saliva | 62.50 (35.56)
  Coughing | 37.40 (30.00)
  Feeling Ill | 21.95 (29.45)
  Painkiller Use | 82.93 (38.09)
  Nutritional Supplement Use | 56.10 (50.24)
  Feeding Tube Use | 58.54 (49.88)
  Weight Loss | 50.00 (50.64)
  Weight Gain | 22.50 (42.29)

13. Secondary Outcome: Quality of Life Using EORTC QLQ-H&N 35 - Cycle 9
Description: as for outcome 11
Time Frame: At Cycle 9 (Week 26)
Population: Treated patients who completed Quality of Life evaluations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reirradiation + MK-3475
Number analyzed (Participants) | 25
score on a scale
  Pain | 29.33 (25.13)
  Swallowing Problems | 31.75 (33.61)
  Sensory Problems | 32.54 (34.35)
  Speech Problems | 40.10 (29.35)
  Trouble with Social Eating | 32.25 (29.97)
  Trouble with Social Contact | 20.27 (26.28)
  Less Sexuality | 32.54 (40.99)
  Teeth Problems | 27.54 (39.76)
  Mouth Opening Problems | 48.00 (43.12)
  Dry Mouth | 52.00 (33.44)
  Sticky Saliva | 52.00 (36.11)
  Coughing | 31.94 (26.88)
  Feeling Ill | 16.00 (29.06)
  Painkiller Use | 68.00 (47.61)
  Nutritional Supplement Use | 62.50 (49.45)
  Feeding Tube Use | 36.00 (48.99)
  Weight Loss | 33.33 (48.15)
  Weight Gain | 16.00 (37.42)

14. Secondary Outcome: Quality of Life Using EORTC QLQ-H&N 35 - 12 Months
Description: as for outcome 11
Time Frame: At 12 months
Population: Treated patients who completed Quality of Life evaluations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reirradiation + MK-3475
Number analyzed (Participants) | 10
score on a scale
  Pain | 10.00 (12.30)
  Swallowing Problems | 52.50 (46.98)
  Sensory Problems | 30.00 (29.19)
  Speech Problems | 51.11 (28.30)
  Trouble with Social Eating | 54.17 (41.99)
  Trouble with Social Contact | 11.33 (16.64)
  Less Sexuality | 33.33 (47.14)
  Teeth Problems | 33.33 (38.49)
  Mouth Opening Problems | 74.07 (36.43)
  Dry Mouth | 66.67 (35.14)
  Sticky Saliva | 46.67 (39.13)
  Coughing | 26.67 (34.43)
  Feeling Ill | 10.00 (22.50)
  Painkiller Use | 60.00 (51.64)
  Nutritional Supplement Use | 80.00 (42.16)
  Feeding Tube Use | 50.00 (52.70)
  Weight Loss | 20.00 (42.16)
  Weight Gain | 10.00 (31.62)

15. Secondary Outcome: Quality of Life Using EORTC QLQ-H&N 35 - 36 Months
Description: as for outcome 11
Time Frame: At 36 months
Population: Treated patients who completed Quality of Life evaluations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reirradiation + MK-3475
Number analyzed (Participants) | 3
score on a scale
  Pain | 0.00 (0.00)
  Swallowing Problems | 66.67 (11.79)
  Sensory Problems | 0.00 (0.00)
  Speech Problems | 59.26 (16.97)
  Trouble with Social Eating | 72.22 (34.69)
  Trouble with Social Contact | 33.33 (57.74)
  Less Sexuality | 33.33 (57.74)
  Teeth Problems | 22.22 (19.25)
  Mouth Opening Problems | 50.00 (23.57)
  Dry Mouth | 33.33 (33.33)
  Sticky Saliva | 44.44 (50.92)
  Coughing | 11.11 (19.25)
  Feeling Ill | 0.00 (0.00)
  Painkiller Use | 33.33 (57.74)
  Nutritional Supplement Use | 100.00 (0.00)
  Feeding Tube Use | 100.00 (0.00)
  Weight Loss | 0.00 (0.00)
  Weight Gain | 0.00 (0.00)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for a total of 6 years, 7 months
Arm/Group | Reirradiation + MK-3475
All-Cause Mortality (participants affected / at risk) | 37/48
Serious Adverse Events (participants affected / at risk) | 27/48
Other Adverse Events (participants affected / at risk) | 46/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reirradiation + MK-3475 (N=48)
Anemia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Death NOS (General disorders) | 3
Fatigue (General disorders) | 2
Fever (General disorders) | 2
Other, specify (General disorders) | 2
Lung infection (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Stoma site infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Injury, poisoning and procedural complications_Fall (Injury, poisoning and procedural complications) | 1
Blood bilirubin increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Weight loss (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reirradiation + MK-3475 (N=48)
Anemia (Blood and lymphatic system disorders) | 16
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 4
Leukocytosis (Blood and lymphatic system disorders) | 2
Cardiac disorders_Palpitations (Cardiac disorders) | 1
Cardiac disorders_Sinus bradycardia (Cardiac disorders) | 2
Cardiac disorders_Sinus tachycardia (Cardiac disorders) | 2
Other, specify (Ear and labyrinth disorders) | 3
Ear pain (Ear and labyrinth disorders) | 7
Hearing impaired (Ear and labyrinth disorders) | 4
Middle ear inflammation (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Hyperthyroidism (Endocrine disorders) | 2
Hypothyroidism (Endocrine disorders) | 9
Blurred vision (Eye disorders) | 2
Eye disorders - Other, specify (Eye disorders) | 3
Photophobia (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 22
Diarrhea (Gastrointestinal disorders) | 10
Dry mouth (Gastrointestinal disorders) | 18
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 16
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 6
Mucositis oral (Gastrointestinal disorders) | 20
Nausea (Gastrointestinal disorders) | 15
Oral hemorrhage (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 13
Salivary duct inflammation (Gastrointestinal disorders) | 3
Stomach pain (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Chills (General disorders) | 1
Edema face (General disorders) | 8
Edema limbs (General disorders) | 5
Facial pain (General disorders) | 3
Fatigue (General disorders) | 32
Fever (General disorders) | 6
Flu like symptoms (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 3
Irritability (General disorders) | 1
Localized edema (General disorders) | 1
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 9
Bile duct stenosis (Hepatobiliary disorders) | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Bladder infection (Infections and infestations) | 1
Bronchial infection (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 6
Lung infection (Infections and infestations) | 2
Mucosal infection (Infections and infestations) | 3
Otitis media (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 1
Scrotal infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 3
Stoma site infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 4
Bruising (Injury, poisoning and procedural complications) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 16
Fall (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 8
Alkaline phosphatase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 9
Cholesterol high (Investigations) | 0
Creatinine increased (Investigations) | 1
GGT increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 7
Lymphocyte count decreased (Investigations) | 11
Platelet count decreased (Investigations) | 1
Weight gain (Investigations) | 1
Weight loss (Investigations) | 21
White blood cell decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 8
Hypercalcemia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 2
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Other, specify (Metabolism and nutrition disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 13
Neck soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 11
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Aphonia (Nervous system disorders) | 2
Ataxia (Nervous system disorders) | 1
Concentration impairment (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 8
Dysarthria (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 9
Headache (Nervous system disorders) | 6
Hypoglossal nerve disorder (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 4
Neuralgia (Nervous system disorders) | 2
Paresthesia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 5
Confusion (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 3
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 5
Proteinuria (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 5
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 6
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 2
Surgical and medical procedures_Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 7
Hypotension (Vascular disorders) | 5
Lymphedema (Vascular disorders) | 2
Other, specify (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/09/NCT02289209/Prot_SAP_000.pdf